CLINICAL TRIAL: NCT01995045
Title: The Effects of Triamcinolone Acetonide With Retrobulbar Anesthesia on Postoperative Pain Control Following Vitreoretinal Surgery
Brief Title: Postoperative Pain Control Following Vitreoretinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Timothy W. Olsen, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00053514
Record Dates: First submitted 2013-11-10; First posted 2013-11-26 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Retinal Detachment; Proliferative Vitreoretinopathy; Retinoschisis
Keywords: Retina; Vitreoretinal; Surgery
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative; Retinoschisis | interventions — Triamcinolone; Triamcinolone Acetonide; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivicaine & Triamcinolone (Experimental): Retrobulbar anesthesia with Bupivicaine Hydrochloride and Triamcinolone Acetonide
  Interventions: Drug: Triamcinolone; Drug: Bupivicaine Hydrochloride
- Bupivicaine (Active Comparator): Retrobulbar anesthesia with Bupivicaine Hydrochloride
  Interventions: Drug: Bupivicaine Hydrochloride

INTERVENTIONS:
Drug: Triamcinolone — Retrobulbar anesthesia
  Other Names: Kenalog; Triamcinolone Acetonide
  Arms: Bupivicaine & Triamcinolone
Drug: Bupivicaine Hydrochloride — Retrobulbar anesthesia
  Other Names: Marcaine

SUMMARY:
The aim of this study is to evaluate if patients receiving a steroid (triamcinolone acetonide) combined with local anesthesia and antibiotic following retina surgery have better postoperative pain control those receiving local anesthesia and antibiotic alone.

DETAILED DESCRIPTION:
Currently, patients undergoing vitreoretinal surgery at the Emory Eye Center and Emory University Hospital receive a injection of local anesthesia behind the eye (retrobulbar) at the start of surgery to minimize discomfort felt during the surgery. At the end of surgery all patients receive a periocular antibiotic and steroid injection. Some patients also receive a retrobulbar injection of local anesthesia (bupivicaine) at the conclusion of surgery in order to decrease postoperative pain and discomfort.

It has been our observation that when the local anesthesia is combined with a steroid (triamcinolone acetonide) in a retrobulbar injection at the conclusion of surgery, patients tend to be pain free for longer intervals then when local anesthesia is used alone. The objective of this study is to evaluate if patients receiving triamcinolone acetonide combined with local anesthesia and antibiotic compared to those receiving local anesthesia and antibiotic alone do better with postoperative pain control.

All eligible patients undergoing vitreoretinal surgery at the Emory Eye Center and Emory University Hospital will be offered enrollment. About 60 patients will be invited to participate in this study. Patients will undergo standard of care surgery. At the conclusion of surgery, patients will receive a retrobulbar antibiotic and anesthetic as standard of care. Half of the patients will receive this mixture plus steroid and the other half will receive this mixture plus saline. On postoperative day 1, patients will be given a questionnaire to assess pain. Pain levels in the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing vitreoretinal surgery at the Emory Eye Center Ambulatory Surgery Center and Emory University Hospital by retina attending faculty surgeons

Exclusion Criteria:

* Unable to verbalize level of pain control
* Pediatric patients (<18 years old)
* Glaucoma, ocular hypertension, or glaucoma suspects
* Allergy to local anesthetic
* Pre-existing chronic pain requiring narcotic pain medication
* Drug addiction
* Impaired periorbital sensation (history of herpes simplex, zoster, corneal graft)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W Olsen, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Eye Center, Atlanta, Georgia, United States

REFERENCES:
- [Background] Gioia L, Prandi E, Codnotti M, Casati A,et al Peribulbar anesthesia with either 0.75% ropivacaine or a 2% lidocaine and 0.5% bupivacaine mixture for vitreoretinal surgery: a double-blinded study. Anesth Analg(89: 739-742, 1999. Shende D, Sadhasivam S, Madan R. Effects of peribulbar bupivacaine as an adjunct to general anaesthesia on peri-operative outcome following retinal detachment surgery. Anaesthesia(55): 970-975, 2000. Morel J, Pascal J, Charier D, et al. Preoperative peribulbar block in patients undergoing retinal detachment surgery under general anesthesia: a randomized double-blind study. Anesth Analg (102): 1082-1087, 2006. Ghali AM, Btarny AM. The effect on outcome of peribulbar anesthesia in conjunction with general anesthesia for vitreoretinal surgery. Anaesthesia (65): 249-253, 2010. Chavan SB, Cummings EJ.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital between October 1, 2012 and June 17, 2016 who were scheduled to have scleral buckle surgery, 20-gauge vitrectomy, or both.
Pre-assignment Details: Of the 58 participants recruited for the study, data for 57 participants were analyzed. Data for one participant was not available for analysis.
Groups:
- Bupivicaine & Triamcinolone: Participants who were scheduled to have scleral buckle surgery, 20-gauge vitrectomy, or both were randomized to receive an injection of a 3-mL mixture of 1 mL 0.75% bupivacaine (7.5 mg/1 mL), 1 mL cefazolin (100mg/mL), and 1 mL triamcinolone (40mg/mL) at the end of surgery.
- Salt Solution, Bupivacaine, and Cefazolin: Participants who were scheduled to have scleral buckle surgery, 20-gauge vitrectomy, or both were randomized to receive an injection of a 3-mL mixture of 1 mL 0.75% bupivacaine (7.5 mg/mL), 1 mL of balanced salt solution (BSS), and 1 mL cefazolin (100mg/mL) at the end of surgery.
Period: Overall Study
Arm/Group | Bupivicaine & Triamcinolone | Salt Solution, Bupivacaine, and Cefazolin
Started | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivicaine & Triamcinolone | Salt Solution, Bupivacaine, and Cefazolin | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 22 | 43
  >=65 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 21 | 20 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Score
Description: The mean pain score assessed by the Visual Analog Pain Scale ranging from 0-10; 10 being the worst possible pain.
Time Frame: Post-Operative Day 1 (Up to 24 hours)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivicaine & Triamcinolone | Salt Solution, Bupivacaine, and Cefazolin
Number analyzed (Participants) | 29 | 28
units on a scale | 2.9 (2.8) | 3.8 (2.8)

2. Secondary Outcome: Mean Acetaminophen Intake
Description: The mean acetaminophen use post surgery in milligrams(mg).
Time Frame: Post Surgery (Up to 24 hours)
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Bupivicaine & Triamcinolone | Salt Solution, Bupivacaine, and Cefazolin
Number analyzed (Participants) | 29 | 28
milligrams | 819 (998) | 962 (839)

3. Secondary Outcome: Mean Hydrocodone Intake
Description: The mean hydrocodone use post surgery in milligrams(mg).
Time Frame: Post Surgery (Up to 24 hours)
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Bupivicaine & Triamcinolone | Salt Solution, Bupivacaine, and Cefazolin
Number analyzed (Participants) | 29 | 28
milligrams | .7 (2.9) | 2.8 (6.0)

4. Secondary Outcome: Mean Oxycodone Intake
Description: The mean oxycodone use post surgery in milligrams(mg).
Time Frame: Post Surgery (Up to 24 hours)
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Bupivicaine & Triamcinolone | Salt Solution, Bupivacaine, and Cefazolin
Number analyzed (Participants) | 29 | 28
milligrams | 6.7 (6.8) | 9.0 (12.9)

ADVERSE EVENTS:
Arm/Group | Bupivicaine & Triamcinolone | Bupivicaine
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 1/29 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivicaine & Triamcinolone (N=29) | Bupivicaine (N=28)
Intraocular Pressure (Eye disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes